CLINICAL TRIAL: NCT05492630
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Ascending Single and Multiple Doses to Evaluate the Safety, Tolerability, Pharmacokinetics/Pharmacodynamics, and Randomized, Open-label, Food Effect Study of HEC73077 in Healthy Subjects
Brief Title: Single and Multiple Dose Safety, Tolerability, PK and Food Effect Study of HEC73077 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC73077-P-01
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HEC73077 tablets (Experimental): Single-Dose Study: There will be a total of 7 dose cohorts. Multiple-dose Study: There will be a total of 4 dose cohorts.
  Interventions: Drug: HEC73077 tablets
- HEC73077 placebo tablets (Placebo Comparator): Single-Dose Study: There will be a total of 7 dose cohorts. Multiple-dose Study: There will be a total of 4 dose cohorts.
  Interventions: Drug: HEC73077 placebo tablets

INTERVENTIONS:
Drug: HEC73077 tablets — Single-Dose Study: Each dose of HEC73077 and placebo will be administered with approximately 240 mL of water in the morning after fasting for at least 10 hours overnight.
  Multiple-dose study:The study doses, administration method (fasted or fed), dosing frequency, and dosing period are all to be determined based on data from the single-dose study and/or multiple-dose study.
  Arms: HEC73077 tablets
Drug: HEC73077 placebo tablets — Single-Dose Study: Each dose of HEC73077 and placebo will be administered with approximately 240 mL of water in the morning after fasting for at least 10 hours overnight.
  Multiple-dose study:The study doses, administration method (fasted or fed), dosing frequency, and dosing period are all to be determined based on data from the single-dose study and/or multiple-dose study.
  Arms: HEC73077 placebo tablets

SUMMARY:
The Safety, Tolerability Pharmacokinetic and Food Effect Study of HEC73077 in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before the trial and fully understand the contents of the trial, the process and possible adverse reactions.
2. Be able to complete the study according to the trail protocol.
3. Subjects (including partners) have no pregnancy plan within 6 months after the last dose of study drug and voluntarily take effective contraceptive measures.
4. subjects and must be 18 to 45 years of age inclusive.
5. Body weight ≥ 45 kg(for female) or ≥ 50 kg(for male) and body mass index（BMI）between 18 and 28 kg / m^2, inclusive, at screening.
6. There was no clinically significant medical history of respiratory, circulatory, digestive, urinary, blood, endocrine, nervous system diseases and metabolic abnormalities at screening.
7. Subjects, who are healthy, as having no clinically significant abnormalities in vital signs, physical examination, clinical laboratory test results, Chest X-ray and 12-lead electrocardiogram (ECG).

Exclusion Criteria:

1. Use of >5 cigarettes per day during the past 3 months.
2. Known history of allergy to study drugs，or allergies constitution ( multiple drug and food allergies).
3. History of alcoholism or drink regularly within 3 months prior to the study (defined as Alcohol consumption of > 14 units/week).
4. Positive results from urine drug screen test.
5. Donation or loss of blood over 450 mL within 3 months prior to screening.
6. Subjects suffering from gastrointestinal diseases that can interfere with absorption or metabolism of drugs within 6 months before screening.
7. Use of any prescription or non-prescription medications within 14 days prior to initial dosing
8. Consume foods or beverages containing caffeine, xanthine, alcohol, and grapefruit within 48 hours prior to initial dosing.
9. Subjects who participated in another clinical trial within 3 months prior to initial dosing.
10. Female subjects were lactating or had positive serum pregnancy results during the screening or testing period.
11. Subjects deemed unsuitable by the investigator for any other reason.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to 19 days
  Incidence of adverse events
Cmax | Day 1-17
  Maximum plasma concentration of study drugs
AUC0-∞ | Day 1-17
  area under the concentration versus time curve (AUC) from time zero to infinity

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China